CLINICAL TRIAL: NCT05194813
Title: The Effect of Surface Treatment of the Dental Implant on the Osseointegration in Mandibular Posterior Missing Teeth
Brief Title: Surface Treatment of the Dental Implant on the Osseointegration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Implants2022
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Dental Implants; Surface Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrophilic sandblasted and acid-etched dental implants (Experimental)
  Interventions: Other: Aqua alvim CM, neodent implant (Test)
- Conventional hydrophobic sandblasted and acid-etched dental implant (Active Comparator)
  Interventions: Other: Neoporous alvim CM, neodent implant (Control)

INTERVENTIONS:
Other: Aqua alvim CM, neodent implant (Test) — Acqua, Hydrophilic sandblasted, and acid-etched dental implants
  Arms: Hydrophilic sandblasted and acid-etched dental implants
Other: Neoporous alvim CM, neodent implant (Control) — Neoporous, Hydrophilic sandblasted, and acid-etched dental implants
  Arms: Conventional hydrophobic sandblasted and acid-etched dental implant

SUMMARY:
Dental implants have become a widely accepted treatment modality for the replacement of missing single or multiple teeth in the recent years. In order to meet patients' needs for shorter treatment times and the necessity of dealing with more challenging clinical situations, implants and implant therapies have undergone continuous improvement to improve the function and longevity of the implants. Recently the constant search for improvements in modern implant have been focused on surface modifications so a new era of surface treatment have been showed up; the chemically modified hydrophilic surfaces.

ELIGIBILITY:
Inclusion Criteria:

* Missing mandibular posterior teeth.
* Good oral hygiene (plaque index less than 10 %)
* Good compliance to the treatment.
* Participants are free from local or systemic disease
* Willingness and ability to commit to follow-up placement.
* Adequate bone height and width to accommodate implant placement and sufficient keratinzed mucosa.
* At least 3months after tooth extraction
* Sufficient interocclusal distance

Exclusion criteria

* Presence of persistent and unresolved infection in the implant site
* Parafunctional habits.
* Heavy Smokers.
* Uncontrolled systemic disease that impedes bone healing

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change in implant stability | at baseline and 6 months
  The implant stability measurement was examined at the time of insertion of the implants (primary stability) and 6 months (secondary stability) for the two groups of patients using the resonance Frequency Analysis (RFA) via the Osstell ISQ system
Change in bone density | at baseline and 6 months
  Cone beam Computerized tomography was used to assess bone denisty
Change in ridge height | at baseline and 6 months
  Cone beam Computerized tomography was used to assess ridge height
Biochemical assessment of bone formation | at 3 months
  Done by measuring of Runt-related transcription factor 2 (RUNX2) as a bone marker by Enzyme-Linked Immunosorbent Assay

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt